CLINICAL TRIAL: NCT04521504
Title: The Use of the Motion Analysis System ISEO, as a Biofeedback Tool During the Rehabilitation Process of Patients Surgically Treated for Rotator Cuff Tear
Brief Title: The ISEO Biofeedback Tool During the Rehabilitation of Patients Treated for Rotator Cuff Tear
Acronym: PDT1-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Collaborators: AUSL Romagna Rimini (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDT1-1
Record Dates: First submitted 2020-08-04; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Rotator Cuff Tears
Keywords: Shoulder; Biofeedback; Kinematics
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: The study considers participants divided in two groups: the control group and the experimental group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback (Experimental): Patients were treated with an experimental rehabilitation protocol, based on shoulder kinematic biofeedback.
  Interventions: Device: Kinematic biofeedback with ISEO motion analysis system
- Control (No Intervention): Patients were treated with a standard rehabilitation protocol, based on hospital guidelines.

INTERVENTIONS:
Device: Kinematic biofeedback with ISEO motion analysis system — Exercises are performed with the help of the ISEO motion analysis system, that provides a real-time biofeedback of shoulder kinematics. All exercises are administered by the Physical Therapist.
  Arms: Biofeedback

SUMMARY:
The present study addresses the issue about post-surgical recovery process, for patients arthroscopically treated for rotator-cuff tear. The aim of the research is to test the effectiveness of a new rehabilitation protocol that includes kinematic biofeedback with the motion analysis system ISEO.

DETAILED DESCRIPTION:
The research includes at least 62 patients arthroscopically treated for the rotator cuff tear. For this purpose, two groups of patients of equal size are identified. The attribution of each patient to one of the two groups is random. The standard rehabilitation protocol is applied to the Control group (Group A), whereas the standard rehabilitation protocol integrated by proprioception exercises (physical therapist assisted) performed with ISEO is applied to the Experimental group (Group B). The primary objective is to verify if the ISEO system, used as a biofeedback tool, improves shoulder functionality and activity of patients arthroscopically treated for rotator cuff tear, both in the short (90 days from surgery) and in the medium term (6-12 months from surgery). All patients are longitudinally evaluated from the pre-surgery to a 6/12 months follow-up. Each evaluation includes both a clinical and an instrumented assessment of shoulder kinematics. The primary outcome tested is the Scapula-Weighted Constant-Murley Score, which represents a reformulation of the Constant-Murley Score, which is modified based on the quality of the scapular movement measured with ISEO.

ELIGIBILITY:
Inclusion Criteria:

* patients with rotator cuff injuries;
* asymptomatic contralateral shoulder, that can be considered as a reference for the differential evaluation;
* indication for arthroscopy;
* employees;
* rehabilitation executed at AUSL-Romagna.

Exclusion Criteria:

* irreparable injuries of the rotator cuff;
* contralateral painful shoulder;
* patients being treated for cancer in the last 6 months;
* patients with concomitant neurological pathologies;
* patients with spinal cord injuries;
* patients with cuff lesions with infectious processes;
* patients with severe scoliosis;
* patients with recurrent lesions of the cuff;
* patients with occupational diseases or work-related accidents;
* patients for whom the return to work cannot be reliably established.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
The Scapula-Weighted Constant-Murley Score (SW-CMS) at T3 | 90 days after surgery
  The SW-CMS is a modified version of the CMS, based on the quality of the movement of the scapula: the score referred to humerus elevation is "weighted" based on scapula movement. The Score varies between 0 (worse) and 100 (best) points.
The Scapula-Weighted Constant-Murley Score (SW-CMS) at T5A | 6 months after surgery
  The SW-CMS is a modified version of the CMS, based on the quality of the movement of the scapula: the score referred to humerus elevation is "weighted" based on scapula movement. The Score varies between 0 (worse) and 100 (best) points.
The Scapula-Weighted Constant-Murley Score (SW-CMS) at T5B | 12 months after surgery
  The SW-CMS is a modified version of the CMS, based on the quality of the movement of the scapula: the score referred to humerus elevation is "weighted" based on scapula movement. The Score varies between 0 (worse) and 100 (best) points.

SECONDARY OUTCOMES:
Constant-Murley Score (CMS) | T0 (before surgery), T1 (45 days after surgery), T3 (90 days after surgery), T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  The CMS is a standard questionnaire for the evaluation of patients with shoulder diseases, one of the most widespread in Europe. The Score varies between 0 (worse) and 100 (best) points.
American Shoulder and Elbow Score (ASES) | T0 (before surgery), T1 (45 days after surgery), T3 (90 days after surgery), T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  The ASES is a very popular questionnaire (in particular in the USA), partly completed from the patient and partly completed from the doctor. The part dedicated to the patient provides for an assessment of pain, instability and daily life activities. The part filled in by the doctor includes 4 items on tenderness. The ASES varies between 0 (worse) and 100 (best) points.
Disabilities of the Arm, Shoulder and Hand (DASH) | T0 (before surgery), T1 (45 days after surgery), T3 (90 days after surgery), T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  The DASH is a very popular questionnaire that quantifies the level of disability of a patient with upper limb disease. The questionnaire is a self-administered by the patient. The DASH varies between 0 (best) and 100 (worse) points.
EuroQol five-dimension scale (EQ-5D) | T0 (before surgery), T1 (45 days after surgery), T3 (90 days after surgery), T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  The EQ-5D is a standard questionnaire for the measure of health outcome. EQ-5D is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The EQ-5D varies between 0 (worse) and 100 (best) points.
Superficial Electromyography (sEMG) | T0 (before surgery), T1 (45 days after surgery), T3 (90 days after surgery), T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  The sEMG is the electrical activity of shoulder superficial muscles. Muscles acquired are: Deltoid (anterior and posterior), Trapezius (upper, medium and lower), Serratus Anterior, Pectoralis Major and Latissimus Dorsi.
Pectoralis Minor length | T0 (before surgery), T1 (45 days after surgery), T3 (90 days after surgery), T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  Pectoralis Minor length in mm
Body Mass Index (BMI) | Before surgery
  The BMI is measure in kg/m^2
Cervical pain: Presence of cervical pain YES or NOT. If YES, why | Before surgery
  It is measured by the Doctor as follows:
  Presence of cervical pain YES or NOT. If YES, why.

OTHER OUTCOMES:
Percent of job-change | T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  Percentage of patients that had to change their job
Degree of satisfaction of the patient: score | T0 (before surgery), T1 (45 days after surgery), T3 (90 days after surgery), T4 (return-to-work time, up to 24 weeks), T5A (6 months after surgery) and T5B (12 months after surgery).
  Evaluation of the satisfaction of the patient during the rehabilitation period. The score varies from 0 (totally unsatisfied) and 10 (totally satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Maria V Filippi, MD, Principal Investigator — AUSL della Romagna; Paolo Paladini, MD, Study Director — AUSL della Romagna; Riccardo Galassi, MD, Study Director — AUSL della Romagna
Locations (1):
- AUSL della Romagna - Cervesi Hospital, Cattolica, Rimini, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parel I, Jaspers E, DE Baets L, Amoresano A, Cutti AG. Motion analysis of the shoulder in adults: kinematics and electromyography for the clinical practice. Eur J Phys Rehabil Med. 2016 Aug;52(4):575-82. Epub 2016 Jul 19. PMID 27434612
- [Background] Cutti AG, Parel I, Pellegrini A, Paladini P, Sacchetti R, Porcellini G, Merolla G. The Constant score and the assessment of scapula dyskinesis: Proposal and assessment of an integrated outcome measure. J Electromyogr Kinesiol. 2016 Aug;29:81-9. doi: 10.1016/j.jelekin.2015.06.011. Epub 2015 Jul 6. PMID 26184668
- [Background] Cutti AG, Parel I, Raggi M, Petracci E, Pellegrini A, Accardo AP, Sacchetti R, Porcellini G. Prediction bands and intervals for the scapulo-humeral coordination based on the Bootstrap and two Gaussian methods. J Biomech. 2014 Mar 21;47(5):1035-44. doi: 10.1016/j.jbiomech.2013.12.028. Epub 2014 Jan 13. PMID 24485513
- [Background] Constant CR, Gerber C, Emery RJ, Sojbjerg JO, Gohlke F, Boileau P. A review of the Constant score: modifications and guidelines for its use. J Shoulder Elbow Surg. 2008 Mar-Apr;17(2):355-61. doi: 10.1016/j.jse.2007.06.022. Epub 2008 Jan 22. No abstract available. PMID 18218327